CLINICAL TRIAL: NCT06428591
Title: Tandem Freedom Feasibility Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-0017517; U1111-1307-6267 (Other: ICTRP)
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1 diabetes; T1D; Tandem; t:slim X2; automated insulin delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Tandem Freedom (Experimental): After a one week run-in period with Control-IQ technology, participants used the Tandem Freedom system for one day with insulin boluses and one day without insulin boluses.
  Participants performed meal and exercise challenges in a supervised hotel setting.
  Interventions: Device: t:slim X2 insulin pump with Tandem Freedom Algorithm

INTERVENTIONS:
Device: t:slim X2 insulin pump with Tandem Freedom Algorithm — Participants will use the Tandem Freedom system for one day with insulin boluses and one day without insulin boluses.

SUMMARY:
This feasibility study is a prospective, single arm study evaluating the Tandem Freedom system in adults with type 1 diabetes. Existing Control-IQ technology users will use Control-IQ technology at home for a 1 week run-in, then will use Tandem Freedom in a supervised hotel setting.

DETAILED DESCRIPTION:
After a 1 week Control-IQ run-in at home, 10 adults who are existing Control-IQ users with type 1 diabetes will use the Tandem Freedom System for 1 day with boluses, and 1 day without boluses, in a supervised hotel setting. Participants will perform meal and exercise challenges. The primary outcome is safety events. CGM time in ranges will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Diagnosis of type 1 diabetes for at least 1 year
* Current Control-IQ user, having been prescribed Control-IQ for at least 3 months
* HbA1c ≤10%, recorded in the last 3 months
* Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol, including performing the weekend hotel observed setting portion of the study.
* Willing to use only aspart (novorapid) or lispro (humalog) insulin with the study pump, with no use of long-acting basal insulin injections, or inhaled insulin with the study pump.
* Have current glucagon product to treat severe hypoglycemia (injectable or nasal) at home (site will provide prescription if they do not have one)

Exclusion Criteria:

* More than 1 episode of diabetic ketoacidosis (DKA) in the past 6 months
* More than 1 episode of severe hypoglycemia (needing assistance) in the past 6 months
* Inpatient psychiatric treatment in the past 6 months
* For Female: Currently pregnant or planning to become pregnant during the time period of study participation

  1. A negative pregnancy test will be required for all females of child-bearing potential
  2. Counseling on appropriate birth control options will be provided to all females of child-bearing potential
* Concurrent use of any non-insulin glucose-lowering agent, other than metformin (for example, GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas).
* Hemophilia or any other bleeding disorder
* Hemoglobinopathy
* History of heart, liver, lung or kidney disease determined by investigator to interfere with the study
* History of allergic reaction to Humalog or Novorapid
* Use of any medications determined by investigator to interfere with study
* Significant chronic kidney disease (which could impact CGM accuracy in investigator's judgment) or hemodialysis
* Concurrent use of any medication that could interfere with the study CGM, such as hydroxyurea
* History of adrenal insufficiency
* History of abnormal TSH consistent with hypothyroidism or hyperthyroidism that is not appropriately treated
* History of gastroparesis
* A condition, which in the opinion of the investigator or designee, would put the participant or study at risk
* Participation in another pharmaceutical or device trial at the time of enrollment or anticipated for during the time period of study participation
* Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc., or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Pinsker, MD, Study Director — Tandem Diabetes Care
Locations (1):
- University of Otago, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten adults with type 1 diabetes (all existing Control-IQ users) were recruited for this study.
Groups:
- Tandem Freedom: After a 1 week Control-IQ run-in, adults with type 1 diabetes will complete a supervised hotel study with the Tandem Freedom system 1 day with boluses, and 1 day without boluses, performing meal and exercise challenges.
Period: Overall Study
Arm/Group | Tandem Freedom
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 10 adults with type 1 diabetes, who were existing users of the t:slim X2 insulin pump with Control-IQ technology for at least 3 months
Groups:
- t:Slim X2 Insulin Pump With Tandem Freedom Algorithm: After a 1 week Control-IQ run-in, adults with type 1 diabetes will complete a supervised hotel study with the Tandem Freedom system 1 day with boluses, and 1 day without boluses, performing meal and exercise challenges.
Arm/Group | t:Slim X2 Insulin Pump With Tandem Freedom Algorithm
Number analyzed (Participants) | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  New Zealand European | 9
  Maori | 1
HbA1c at Enrollment [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 6.8 (0.7)
Total Daily Insulin Dose at Enrollment [Mean (Standard Deviation); unit: units/day] | 62.3 (22.7)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 18.1 (12.5)
BMI at Enrollment [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (5.8)
Number of DKA events in the last 6 months [Number; unit: DKA events] | 0
Number of severe hypoglycemic events (required assistance) in the last 6 months [Number; unit: Severe Hypoglycemic Events] | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (19.6)

OUTCOME MEASURES:

1. Primary Outcome: Severe Hypoglycemia Events
Description: Number of severe hypoglycemia events (with cognitive impairment such that assistance of another individual is needed for treatment)
Time Frame: Control-IQ Run-in with boluses 7 days, day 8 freedom with meal bolus and day 9 freedom without meal bolus
Measure: Number; unit: number of events
Arm/Group | t:slim X2 insulin pump with Tandem Freedom Algorithm
Number analyzed (Participants) | 10
number of events
  Control-IQ Run-In with Boluses (7 Days) | 0
  Freedom with Meal Boluses (24 Hours) | 0
  Freedom without Meal Boluses (24 Hours) | 0

2. Primary Outcome: Diabetic Ketoacidosis Events
Description: Number of diabetic ketoacidosis events
Time Frame: Control-IQ Run-in with boluses 7 days, day 8 freedom with meal bolus and day 9 freedom without meal bolus
Measure: Number; unit: number of events
Arm/Group | t:slim X2 insulin pump with Tandem Freedom Algorithm
Number analyzed (Participants) | 10
number of events
  Control-IQ Run-In with Boluses (7 Days) | 0
  Freedom with Meal Boluses (24 Hours) | 0
  Freedom without Meal Boluses (24 Hours) | 0

3. Secondary Outcome: Percent Time <54 mg/dL
Description: CGM measured percent time <54 mg/dL
Time Frame: Control-IQ Run-in with boluses 7 days, day 8 freedom with meal bolus and day 9 freedom without meal bolus
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
percentage of time
  Control-IQ Run-In with Boluses (7 Days) | 0.1 [0.0 to 0.3]
  Freedom with Meal Boluses (24 Hours) | 0.0 [0.0 to 0.3]
  Freedom without Meal Boluses (24 Hours) | 0.0 [0.0 to 0.0]

4. Secondary Outcome: Percent Time <70 mg/dL
Description: CGM measured percent time <70 mg/dL
Time Frame: Control-IQ Run-in with boluses 7 days, day 8 freedom with meal bolus and day 9 freedom without meal bolus
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | t:slim X2 insulin pump with Tandem Freedom Algorithm
Number analyzed (Participants) | 10
percentage of time
  Control-IQ Run-In with Boluses (7 Days) | 1.3 [1.1 to 1.8]
  Freedom with Meal Boluses (24 Hours) | 1.4 [0.0 to 5.1]
  Freedom without Meal Boluses (24 Hours) | 0.0 [0.0 to 1.3]

5. Secondary Outcome: Percent Time in Range 70 - 180 mg/dL
Description: CGM measured percent time in range 70 - 180 mg/dL
Time Frame: Control-IQ Run-in with boluses 7 days, day 8 freedom with meal bolus and day 9 freedom without meal bolus
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
percentage of time
  Control-IQ Run-In with Boluses (7 Days) | 61.8 [56.0 to 72.8]
  Freedom with Boluses (24 Hours) | 82.4 [52.2 to 86.5]
  Freedom without Boluses (24 Hours) | 54.7 [47.1 to 73.7]

6. Secondary Outcome: Percent Time in Range 70 - 140 mg/dL
Description: CGM measured percent time in range 70 - 140 mg/dL
Time Frame: Control-IQ Run-in with boluses 7 days, day 8 freedom with meal bolus and day 9 freedom without meal bolus
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
percentage of time
  Control-IQ Run-In with Boluses (7 Days) | 37.2 [30.1 to 49.8]
  Freedom with Boluses (24 Hours) | 46.5 [26.1 to 60.8]
  Freedom without Boluses (24 Hours) | 34.7 [25.7 to 37.8]

7. Secondary Outcome: Percent Time >180 mg/dL
Description: CGM measured percent time >180 mg/dL
Time Frame: Control-IQ Run-in with boluses 7 days, day 8 freedom with meal bolus and day 9 freedom without meal bolus
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
percentage of time
  Control-IQ Run-In with Boluses (7 Days) | 36.9 [25.5 to 43.0]
  Freedom with Meal Boluses (24 Hours) | 13.5 [9.3 to 46.2]
  Freedom without Meal Boluses (24 Hours) | 44.4 [26.3 to 51.9]

8. Secondary Outcome: Percent Time >250 mg/dL
Description: CGM measured percent time >250mg/dL
Time Frame: Control-IQ Run-in with boluses 7 days, day 8 freedom with meal bolus and day 9 freedom without meal bolus
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
percentage of time
  Control-IQ Run-In with Boluses (7 Days) | 9.1 [5.2 to 15.2]
  Freedom with Meal Boluses (24 Hours) | 0.0 [0.0 to 12.4]
  Freedom without Meal Boluses (24 Hours) | 3.5 [1.4 to 11.5]

9. Secondary Outcome: Mean Glucose (mg/dL)
Description: CGM measured mean glucose (mg/dL)
Time Frame: Control-IQ Run-in with boluses 7 days, day 8 freedom with meal bolus and day 9 freedom without meal bolus
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
mg/dL
  Control-IQ Run-In with Boluses (7 Days) | 170.6 [151.3 to 176.7]
  Freedom with Meal Boluses (24 Hours) | 139.6 [127.2 to 180.5]
  Freedom without Meal Boluses (24 Hours) | 175.6 [151.5 to 182.2]

10. Secondary Outcome: Glucose Coefficient of Variation (%)
Description: CGM measured Coefficient of Variation (%)
Time Frame: Control-IQ Run-in with boluses 7 days, day 8 freedom with meal bolus and day 9 freedom without meal bolus
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
percentage
  Control-IQ Run-In with Boluses (7 Days) | 35.9 [34.4 to 37.6]
  Freedom with Meal Boluses (24 Hours) | 29.1 [22.0 to 32.5]
  Freedom without Meal Boluses (24 Hours) | 27.4 [25.7 to 30.1]

11. Secondary Outcome: Glucose Standard Deviation (mg/dL)
Description: CGM measured Standard Deviation (mg/dL)
Time Frame: Control-IQ Run-in with boluses 7 days, day 8 freedom with meal bolus and day 9 freedom without meal bolus
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
mg/dL
  Control-IQ Run-In with Boluses (7 Days) | 59.6 [51.3 to 67.2]
  Freedom with Meal Boluses (24 Hours) | 37.1 [29.0 to 61.6]
  Freedom without Meal Boluses (24 Hours) | 44.4 [42.0 to 49.6]

ADVERSE EVENTS:
Time Frame: 9 days, to include a 7 day run-in with Control-IQ technology, followed by one day of Freedom with boluses and one day of Freedom without boluses.
Arm/Group | t:slim X2 insulin pump with Tandem Freedom Algorithm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | t:slim X2 insulin pump with Tandem Freedom Algorithm (N=10)
Hyperglycemia with ketosis, due to infusion set failure (Endocrine disorders) | 1 (1) — While using Freedom with boluses, resolved with infusion set change.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT06428591/Prot_SAP_000.pdf